CLINICAL TRIAL: NCT05173311
Title: Pilot Study: The Effectiveness of a Mobile Application in Increasing Vegetable Acceptance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: University of Warsaw (Other); University of Eastern Finland (Other); Folkhälsan Research Center (Unknown); Tampere University (Other); EIT Food (Unknown)
Responsible Party: Principal Investigator, Henna Vepsalainen, Principal investigator, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19057
Record Dates: First submitted 2021-11-29; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Healthy Nutrition; Eating Behavior
Keywords: Games for health; Mobile application; Smartphone application; Randomized trial
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application use arm (Experimental): The early childhood education and care (ECEC) professionals in the intervention arm groups were instructed to use the application with a tablet computer at least 1-2 times a week during the intervention period (3-4 weeks) and to record the number of tasks completed by their group in a logbook. In addition, we recommended that each group focus on at least six vegetables or fruits during the intervention period.
  Interventions: Behavioral: Intervention arm
- Control arm (No Intervention): The control arm groups were instructed to continue their normal routines during the intervention period. They were instructed to refrain from introducing any novel food education methods during the intervention period.

INTERVENTIONS:
Behavioral: Intervention arm — The intervention arm groups were instructed to use the Mole's Veggie Adventures mobile application for 3-4 weeks.
  Other Names: Mole's Veggie Adventures
  Arms: Application use arm

SUMMARY:
The purpose of this study was to examine the effectiveness of the Mole's Veggie Adventures mobile application in increasing fruit and vegetable acceptance among 3-6-year-olds.

DETAILED DESCRIPTION:
After the parents of the participating children had signed an informed consent and filled in the baseline questionnaires, the participating early childhood education and care (ECEC) centers (in Finland) or groups within the ECEC centers (in Poland) were randomly allocated into intervention and control arms. Researchers visited the intervention arm groups and introduced the application to the ECEC professionals. The ECEC professionals were instructed to use the application with a tablet computer at least one to two times a week during the intervention period (3-4 weeks) and to record the number of tasks completed by their group in a logbook. In addition, the research team recommended that each group focuses on at least six vegetables or fruits during the intervention period. The control arm groups were instructed to continue their normal routines during the intervention period and to refrain from introducing any novel food education methods during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* All children in the participating early childhood education and care (ECEC) groups

Exclusion Criteria:

* None

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 326 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Fruit and vegetable acceptance (post intervention) | The parents filled in the questionnaire after the intervention (4-5 weeks after the onset of the intervention).
  The parents filled in a questionnaire listing 25 vegetables and fruits and inquiring whether these had been offered to the child during the past 4 weeks and how the child reacted to those that had been served. All the listed vegetables and fruits were introduced in the app. The answer options were 0=was not offered during the past four weeks, 1=refused to touch food, 2=touched food but did not put in/near mouth, 3=put food to lips but not in mouth, 4=put food in mouth but spat out/did not eat, and 5=ate food. For each participant, we calculated an fruit and vegetable acceptance score by summing the answers to each of the 25 vegetable and fruit items, with higher scores indicating a higher fruit and vegetable acceptance (theoretical range 0-125).
Relative fruit and vegetable acceptance (post intervention) | The parents filled in the questionnaire after the intervention (4-5 weeks after the onset of the intervention).
  Using the same questionnaire, we calculated the number of fruits and vegetables served during the past 4 weeks (range 0-25) and used this information to create a relative fruits and vegetable acceptance score (range 0-5) by dividing the fruits and vegetable acceptance score by the number of fruits and vegetables served.

SECONDARY OUTCOMES:
Emotionality (post intervention) | The parents filled in the questionnaire after the intervention (4-5 weeks after the onset of the intervention).
  The parents filled in a questionnaire describing the emotionality of the children using a Likert scale (1-5). The questionnaire covered four emotions. An average of two items per emotion were used to calculate the variables (scale 1-5).
Emotion regulation (post intervention) | The parents filled in the questionnaire after the intervention (4-5 weeks after the onset of the intervention).
  The parents filled in a questionnaire describing the emotion regulation of the children using a Likert scale (1-5). The questionnaire covered four emotions. An average of two items per emotion were used to calculate the variables (scale 1-5).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vepsalainen H, Skaffari E, Wojtkowska K, Barlinska J, Kinnunen S, Makkonen R, Heikkila M, Lehtovirta M, Ray C, Suhonen E, Nevalainen J, Sajaniemi N, Erkkola M. A Mobile App to Increase Fruit and Vegetable Acceptance Among Finnish and Polish Preschoolers: Randomized Trial. JMIR Mhealth Uhealth. 2022 Jan 4;10(1):e30352. doi: 10.2196/30352. PMID 34982718
- See also: A video demonstrating the most important sections of the current version of the Mole's Veggie Adventures application. — https://www.youtube.com/watch?v=c5XXH-C-LhA